CLINICAL TRIAL: NCT05645458
Title: The Effect of the Mobile Application for Caregivers of Patients With Percutaneous Endoscopic Gastrostomy (PEG) on the Competence, Satisfaction and Care Burden of Caregivers
Brief Title: The Effect of the Mobile Application for Caregivers of Patients With Percutaneous Endoscopic Gastrostomy (PEG) on Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: duzceUatiye-3
Record Dates: First submitted 2022-12-02; First posted 2022-12-09 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Percutaneous Endoscopic Gastrostomy; Caregiver Burden; Mobile Application
Keywords: mobile application; Percutaneous endoscopic gastrostomy; caregiver burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Pre-tests will be applied to the caregiver before the patient is discharged, and the first data will be obtained by observing during PEG care. Then, traditional training on PEG care will be given to the patient's relatives. The tests applied after this training will be applied again. Tests and observation forms will be applied in the 1st month and 3rd month after discharge. By making home visit the participant, recording will be video-recorded so that his identity will not be seen while he is doing PEG care, and the recording will be transcribed to the observation form by 2 blinded people other than the researcher.
- experimental group (Experimental): In addition to maintaining the control group, the experimental group is monitored by installing the mobile application we have developed.
  Interventions: Other: mobile application ( PEG Assist )

INTERVENTIONS:
Other: mobile application ( PEG Assist ) — The mobile application is used for PEG care. İt gives some information to caregivers related to PEG, PEG care, etc. Also, the researcher can monitor all feeding times with this application.
  Arms: experimental group

SUMMARY:
• Brief Summary: In order to benefit from the opportunity of education anytime and anywhere with distance education, individuals need to use mobile devices such as mobile phones, tablets, PCs, which provide the opportunity to access educational content independent of time and place. For these reasons, new searches for the delivery of health services are on the agenda and mobile health applications are seen as a solution to most problems faced by the health system and hospitals.

Percutaneous endoscopic gastrostomy (PEG) is a nutritional method that was first described by Gauder et al. in 1980 and is used in patients with impaired oral intake and intact gastrointestinal tract for various reasons. Caregivers play an important role in the home care process of patients undergoing PEG. Caregivers may encounter social, physical and psychological problems while applying their care. In line with all these reasons, the training to be given to the patient or his/her relative/person who will perform the PEG implantation is very important.

Aim: The aim of this study is to evaluate the effect of mobile application use in training given to caregivers of patients with PEG on the competence, satisfaction and care burden of caregivers.

DETAILED DESCRIPTION:
Method: Pre-tests will be applied to the caregiver before the patient is discharged, and the first data will be obtained by observing during PEG care. Then, traditional training on PEG care will be given to the relatives of the patients. The tests applied after this training will be applied again.

Your assignments to the research groups that will be formed after the training will be randomly assigned. In this method, which group you will be in will be determined by the computer with the random assignment method. In the experimental design of the research, a random design with a pretest-posttest control group will be applied. The data obtained will be evaluated with intention-to-treat analysis in case of death of the patient who stopped working for any reason after starting the research, started feeding with a method other than PEG, or was cared for.After randomization, the participant in the experimental group will be taught to use the mobile application by the researcher. Tests and observation form will be applied to both groups in the 1st and 3rd months after discharge. By making a home visit to the participant, the recording will be video-recorded so that his identity will not be seen while he is doing PEG care, and the recording will be transcribed to the observation form by 2 blinded people other than the researcher. In the experimental design of the research, a random design with pretest-posttest control group will be applied. In our study, all initiatives except the mobile application were designed to be the same in both groups.

Data accumulation methods:

* Mobile app usability scale, Mobile app usage loyalty scale and app use willingness scale
* Mobile application evaluation form
* PEG care competency form
* Maintenance load scale
* Percutaneous Endoscopic Gastrostomy (PEG) Care Observation Form Mobile application: There are two different types of users in the mobile application we have developed. The first user is the user who manages the application and will see the statistics of the entered data. The second user is the user who will provide data entry to the application and care for the patient. After the caregiver downloads and logs in the application, they will be able to save and use the information about their patient. In our application, there is a panel with general information and panels on nutrition, drug administration and stoma care. Caregivers will be able to access information and videos by entering here. In addition, the application will be able to remind some situations such as feeding times by sending notifications according to the patient data entered at the beginning. Apart from these, the thought and caregivers who have a platform where they can consult the nurse will be able to consult the assistant researcher when something is on their minds.

ELIGIBILITY:
Inclusion Criteria:

* Being the first to care for a patient with PEG at Kocaeli State Hospital or Kocaeli University Hospital
* Be able to read and write
* Not have any physical or psychological disability
* Being able to use a mobile application compatible phone or tablet
* Volunteering to work

Exclusion Criteria:

* The patient to be cared for has metastatic cancer
* Refusing to participate in the study
* Stop working at any stage of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Caregiver burden | one day
  The Zarit Caregiver Burden Scale is used to measure caregiver burden. The scale, which is used to determine the effect of caregiving on the individual's life, can be filled by the caregivers themselves or the researcher. It is a five-point Likert type (0 = never, 4 = almost always) and consists of 22 statements. Evaluation of ZBYS is made over the total score. The higher the score, the higher the care burden. A minimum of 0 and a maximum of 88 points are obtained from the scale. Received points; It is evaluated by grading as (0-20) little/no load, (21-40) moderate load, (41-60) severe load, and (61-88) overload.
competence of caregivers | one day
  We use two different form to measure caregiver competence.
  First form is an observation form : This form include was developed by researcher. The participants will be video-recorded in a way that their identity will not be seen while they are doing percutaneous endoscopic gastrostomy care by making a home visit, and the recording will be transcripted to the observation form prepared by the researcher (by 2 people who were blinded except the researcher).
  the second form is the information form: we use this form to measure the information level of the caregiver. this form includes 25 questions related to PEG care. We will compare all participants according to total scores.

SECONDARY OUTCOMES:
Mobile application satisfaction | one day
  We use two different forms to measure mobile application satisfaction level
  The first form satisfaction form was created by the researchers in the form of 4 open-ended questions in order to determine the satisfaction of the mobile application user with the application.
  The second form measures mobile application usability. We will use the Mobile application usability scale/ Mobile application usage loyalty scale and mobile application usage willingness scale developed by Hoehle, Aljafari (2016) et al. Turkish validity and reliability of the scales developed by Güler (2019). The scales are 7-point Likert type and the mobile application usability scale consists of 40 items in total with 10 factors, the Mobile Application Usage Loyalty scale consists of a total of 5 items with a single factor, and the mobile application willingness to use scale consists of 6 items with a single facto

CONTACTS AND LOCATIONS:
Overall Officials: Atiye Erbaş, PhD, Principal Investigator — Duzce University
Locations (1):
- Kocaeli State Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No